CLINICAL TRIAL: NCT03750955
Title: Induced Gingivitis & Intra-oral Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Richard Darveau, Professor, School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SITE00000993
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Plaque Induced Gingivitis

STUDY DESIGN:
Intervention Model Description: Split-mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Plaque induced gingivitis (Experimental): Non-invasive microimaging (OTC device) of gingival tissue where plaque induced gingivitis results from a cessation of oral hygiene in a sextant using a stent-induced biofilm overgrowth model.
  Interventions: Device: Plaque induced gingivitis
- Oral hygiene maintenance (Active Comparator): Non-invasive microimaging (OTC device) of gingival tissue where oral hygiene (tooth brushing with fluoride toothpaste and flossing twice daily) is maintained.
  Interventions: Device: Oral hygiene maintenance

INTERVENTIONS:
Device: Plaque induced gingivitis — Non-invasive microimaging (OTC device) of gingival tissue where oral hygiene cessation utilizing localized stent-induced biofilm overgrowth model (SIBO), will manipulate the participants' oral environment by leading to reversible inflammation of the gingival tissues.
  Other Names: Cessation of oral hygiene
  Arms: Plaque induced gingivitis
Device: Oral hygiene maintenance — Non-invasive microimaging (OTC device) of gingival tissue where oral hygiene has been maintained by tooth brushing with fluoride toothpaste and flossing twice daily.
  Arms: Oral hygiene maintenance

SUMMARY:
Using an experimental, non-invasive intra-oral imaging device, this study evaluates the effects on the gingival tissue when oral hygiene is stopped in a section of the mouth for two weeks and gingivitis develops. The effects on the gingival tissue continues to be evaluated as oral hygiene is resumed and the gingival tissue returns to health.

DETAILED DESCRIPTION:
The study will include the following phases - 1) Hygiene phase of 2 weeks; 2) Gingivitis induction phase with stent lasting up to 2 weeks; and 3) Resolution phase of 2 weeks.

The intervention will consist of cessation of oral hygiene versus an active control of oral hygiene with a fluoridated toothpaste. This study is a modification of classical experimental gingivitis model. The study will prospectively enroll subjects and assign a maxillary sextant to the intervention, while the other sextant will serve as control in a split-mouth design of localized experimental gingivitis, utilizing localized stent-induced biofilm overgrowth model (SIBO). The intervention, i.e. oral hygiene cessation will manipulate the participants' oral environment by leading to reversible inflammation of the gingival tissues. The purpose of this study is to evaluate the effects of oral hygiene cessation in the gingival tissues by an innovative non-invasive microimaging technique, i.e. Optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* In good general health, ASA I
* No clinical signs of gingival inflammation at >90% sites observed
* Probing Depth(PD) ≤ 3.0 mm
* Attachment Loss (AL) = 0 mm
* Gingival health at baseline visit (Day 0): Gingival Index (GI) ≤ 0.5, Bleeding on probing (BOP)(-)
* Fluent in English

Exclusion Criteria:

* • Medical condition which requires premedication prior to dental treatments/visits

  * Subjects unable or unwilling to undergo informed consent process.
  * Subjects currently using anti-gingivitis oral rinses (washout period of 1 week)
  * History of periodontal disease
  * History of systemic inflammatory or immune conditions
  * Use of antibiotic or anti-inflammatory drugs within 30 days of enrollment
  * Pregnant or breastfeeding at time of screening
  * Concurrent orthodontic treatment
  * Untreated carious lesions and/or inadequate restorations, implants, crowns on maxillary non-molar teeth
  * Participation in any other clinical study or test panel within 1 week prior to enrollment into this study
  * Use of tobacco products
  * Subjects who must receive dental treatment during the study dates
  * Orthodontic bands, appliances, or crowns and bridges, or removable partial dentures affecting the non-molar maxillary teeth
  * Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Darveau, MS, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Dentistry, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: L(left) or R(right) maxillary sextant
Groups:
- Plaque Induced Gingivitis: Plaque induced gingivitis resulting from a cessation of oral hygiene in maxillary sextant right (teeth #5 to #8) or left (#9 to #12) using a stent-induced biofilm overgrowth (SIBO) model.
- Oral Hygiene Maintenance: Oral hygiene (tooth brushing with fluoride toothpaste and flossing twice daily) is maintained in a maxillary right (teeth #5 to #8) or left (#9 to #12) sextant.
Period: Hygiene Phase of 2 Weeks
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Started | 16; 16 L(left) or R(right) maxillary sextant (No intervention during the hygiene phase.) | 16; 16 L(left) or R(right) maxillary sextant (No intervention during the hygiene phase.)
Completed | 13; 13 L(left) or R(right) maxillary sextant | 13; 13 L(left) or R(right) maxillary sextant
Not Completed | 3; 3 L(left) or R(right) maxillary sextant | 3; 3 L(left) or R(right) maxillary sextant
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Not eligible at Baseline (start of gingivitis induction phase) | 1 | 1
Period: Gingivitis Induction Phase of 2 Weeks
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Started | 13; 13 L(left) or R(right) maxillary sextant | 13; 13 L(left) or R(right) maxillary sextant
Completed | 13; 13 L(left) or R(right) maxillary sextant (6 participants randomized to L maxillary sextant SIBO; 7 randomized to R maxillary sextant SIBO.) | 13; 13 L(left) or R(right) maxillary sextant (6 randomized to R max. sextant oral hygiene maintenance (OHM); 7 randomized to L max. sextant OHM.)
Not Completed | 0; 0 L(left) or R(right) maxillary sextant | 0; 0 L(left) or R(right) maxillary sextant
Period: Resolution Phase of 2 Weeks
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Started | 13; 13 L(left) or R(right) maxillary sextant (No stent in use; oral hygiene resumed.) | 13; 13 L(left) or R(right) maxillary sextant (Oral hygiene maintenance continued.)
Completed | 13; 13 L(left) or R(right) maxillary sextant | 13; 13 L(left) or R(right) maxillary sextant
Not Completed | 0; 0 L(left) or R(right) maxillary sextant | 0; 0 L(left) or R(right) maxillary sextant

BASELINE CHARACTERISTICS:
Units Other Than Participants: L(left) and R(right) Maxillary sextant
Groups:
- Plaque Induced Gingivitis: Plaque induced gingivitis resulting from a cessation of oral hygiene in a maxillary right (teeth #5 to #8) or left (#9 to #12) sextant using a stent-induced biofilm overgrowth model.
- Total: Total of all reporting groups
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance | Total
Number analyzed (Participants) | 13 | 13 | 13
Number analyzed (L(left) and R(right) Maxillary sextant) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 23.3 [20 to 33] | 23.3 [20 to 33] | 23.3 [20 to 33]
Sex/Gender, Customized [Number; unit: participants]
  Female | 7 | 7 | 7
  Male | 6 | 6 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native, Hispanic or Latino | 0 | 0 | 0
  American Indian or Alaska Native, Not Hispanic or Latino | 0 | 0 | 0
  Asian, Hispanic or Latino | 0 | 0 | 0
  Asian, Not Hispanic or Latino | 8 | 8 | 8
  Native Hawaiian or Other Pacific Islander, Hispanic or Latino | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander, Not Hispanic or Latino | 0 | 0 | 0
  Black or African American, Hispanic or Latino | 0 | 0 | 0
  Black or African American, Not Hispanic or Latino | 0 | 0 | 0
  White, Hispanic or Latino | 1 | 1 | 1
  White, Not Hispanic or Latino | 1 | 1 | 1
  More than one race, Hispanic or Latino | 0 | 0 | 0
  More than one race, Not Hispanic or Latino | 2 | 2 | 2
  Unknown or Not Reported, Hispanic or Latino | 1 | 1 | 1
  Unknown or Not Reported, Not Hispanic or Latino | 0 | 0 | 0
Gingival Index [Mean (Standard Deviation); unit: units on a scale] — Loe and Silness Gingival Index (GI); scale: 0 = normal gingiva, 1 = mild inflammation, 2 = moderate inflammation, 3 = severe inflammation
  units on a scale | 0.085 (0.3) | 0.055 (0.3) | 0.077 (0.12)
Visible Plaque Index [Mean (Standard Deviation); unit: units on a scale] — Scoring: 0 = no plaque; 1 = visible plaque
  units on a scale | 0.078 (0.3) | 0.05 (0.2) | 0.067 (0.12)
Angiogenesis chemokine - angiopoietin-1 [Mean (Standard Deviation); unit: picograms/milliliter] | 141213.37 (338487.23) | 165053.91 (408314.93) | 153133.62 (367653.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Gingivitis at Day 14 as Measured by Non-invasive Microimaging and Gingival Index.
Description: The predictive validity of a non-invasive microimaging technique for assessing experimental gingivitis (plaque induced), as compared with gingival index is not reported. The microimaging technique was used to measure changes in the gingival thickness of the inter-dental tooth area. This area measured did not represent the clinical status of the tissue surrounding the tooth.
  The gingival index is reported. Loe and Silness Gingival Index (GI); scale: 0 = normal gingiva, 1 = mild inflammation, 2 = moderate inflammation, 3 = severe inflammation
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Number analyzed (Participants) | 13 | 13
units on a scale | 0.6 (1.2) | 0.15 (0.3)

2. Primary Outcome: Change From Day 14 Gingivitis at Day 28 as Measured by Non-invasive Microimaging and Gingival Index.
Description: as for outcome 1
Time Frame: Day 14 to Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Number analyzed (Participants) | 13 | 13
units on a scale | 0.08 (0.4) | 0.08 (0.2)

3. Secondary Outcome: Change From Baseline Gingivitis at Day 14 as Measured by Non-invasive Microimaging and Plaque Index.
Description: The predictive validity of a microimaging technique for assessing experimental gingivitis, as compared with plaque index is not reported. The microimaging technique was used to measure changes in the gingival thickness of the inter-dental tooth area. This area measured did not represent the clinical status of the tissue surrounding the tooth.
  The plaque index is reported. Visible Plaque Index; scoring: 0 = no plaque; 1 = visible plaque
Time Frame: Baseline to Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Number analyzed (Participants) | 13 | 13
units on a scale | 0.84 (1.4) | 0.17 (0.24)

4. Secondary Outcome: Change From Day 14 Gingivitis at Day 28 as Measured by Non-invasive Microimaging and Plaque Index.
Description: as for outcome 3
Time Frame: Day 14 to Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Number analyzed (Participants) | 13 | 13
units on a scale | 0.11 (0.18) | 0.105 (0.5)

5. Secondary Outcome: Change From Baseline Angiogenesis Chemokine Concentration at Day 28
Description: Assessment of the concentration of the angiogenesis chemokine angiopoietin-1 during experimental gingivitis.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance
Number analyzed (Participants) | 13 | 13
picograms/milliliter | 137825.56 (339893.64) | 164411.80 (408590.49)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants were questioned at each visit about adverse events since the previous visit.
Groups:
- Hygiene Phase: Adverse Events that occurred during the Hygiene Phase of 2 weeks (the period between enrollment and the start of the Gingivitis Induction Phase of 2 weeks).
- Systemic Adverse Events: Adverse Events that occurred during the Gingivitis Induction Phase of 2 weeks and the Resolution Phase 2 weeks but are not specifically attributable to either the Plaque Induced Gingivitis intervention or the Oral Hygiene Maintenance intervention as the two interventions occurred simultaneously in each participant.
Arm/Group | Plaque Induced Gingivitis | Oral Hygiene Maintenance | Hygiene Phase | Systemic Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 4/13 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plaque Induced Gingivitis (N=13) | Oral Hygiene Maintenance (N=13) | Hygiene Phase (N=13) | Systemic Adverse Events (N=13)
rhinorrhea (Infections and infestations) | 0 | 0 | 1 | 0
menstrual cramps (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
cold (Infections and infestations) | 0 | 0 | 0 | 1
ulcerated interdental papilla #14/15 (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
bruised achilles tendon (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
abraded palatal tissue left posterior (Gastrointestinal disorders) | 0 | 0 | 0 | 1
tender maxillary left posterior buccal gingiva (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03750955/Prot_SAP_000.pdf